CLINICAL TRIAL: NCT06825091
Title: Is Adaptive SBRT for Prostate vs Image-guided Radiotherapy a True Evolution (ASPIRE)
Acronym: ASPIRE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-5757
Record Dates: First submitted 2025-01-26; First posted 2025-02-13 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Localized Prostate Cancer; Stereotactic Body Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-adaptive image-guided SBRT (Other): Patients will receive prostate SBRT. A dose of either 36.25 Gy in 5 fractions (per PACE-B trial) or 42.7 Gy in 7 fractions (per HYPO-RT-PC trial) will be prescribed as per standard practice at PMH. Patients will receive SBRT every other day, excluding weekends and holidays, as per standard practice. Patients will undergo radiotherapy simulation as per standard practice with CT and MR simulation (or without MR if contraindication).
  Interventions: Radiation: SBRT
- Adaptive SBRT (Other): Patients will receive prostate SBRT. A dose of either 36.25 Gy in 5 fractions (per PACE-B trial) or 42.7 Gy in 7 fractions (per HYPO-RT-PC trial) will be prescribed as per standard practice. Patients will receive SBRT every other day, excluding weekends and holidays, as per standard practice. Patients will undergo radiotherapy simulation as per standard practice with CT and MR simulation (or without MR if contraindication).
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Standard of care SBRT (36.25 Gy in 5 fractions or 42.7 Gy in 7 fractions) for localized prostate cancer, delivered either via an adaptive or a non-adaptive image-guided treatment. Androgen deprivation therapy use and duration is at the discretion of the treating physician and patient, in accordance with standard practice based on patients' prostate cancer risk group.

SUMMARY:
The ASPIRE study is a Phase III randomized, single-center study designed to evaluate whether adaptive stereotactic body radiotherapy (SBRT) offers superior clinical benefits compared to standard image-guided SBRT for patients with localized prostate cancer. It aims to explore whether adaptive SBRT can improve urinary outcomes while maintaining effective cancer control.

This interventional study is randomized, single-institution, and includes 320 participants with localized prostate cancer. Patients will be stratified based on fractionation schedules (5 vs. 7 fractions), use of rectal spacers, androgen deprivation therapy (ADT), and baseline alpha receptor antagonist use. Participants will be randomized to receive either adaptive SBRT or standard image-guided SBRT, with both arms adhering to established dosing protocols.

Inclusion criteria includes an age greater than 18 years, diagnosed with localized prostate adenocarcinoma, and an ECOG performance status of 0-1, Eligible for prostate SBRT. The exclusion criteria includes patients who plan for elective nodal irradiation and contraindications to radiotherapy or MRI (for MR-Linac patients).

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Histologic diagnosis of prostate adenocarcinoma
3. Localized prostate cancer
4. Low risk, intermediate risk, or high risk allowed
5. Patient planned for prostate SBRT

Exclusion Criteria:

1. Planned for elective nodal irradiation
2. Contraindications to radiotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2030-02-04 (Estimated); Study Completion 2030-02-04 (Estimated)

PRIMARY OUTCOMES:
To determine whether adaptive SBRT can significantly reduce the proportion of patients experiencing a minimal clinically important difference in patient reported urinary domain changes when compared to the non adaptive image guided SBRT group. | Within 3 months following radiation therapy
  To determine whether adaptive SBRT can significantly reduce the proportion of patients experiencing a minimal clinically important difference (MCID; defined as >10-point change) in patient reported urinary domain changes by EPIC-26 (The Expanded Prostate Cancer Index Composite) questionnaire. within 3-months following radiation when compared to the non-adaptive image guided SBRT group

SECONDARY OUTCOMES:
To determine whether adaptive SBRT to prostate compared to non adaptive image guided SBRT to prostate results in different rates of patient reported outcomes, acute toxicity. | Within 3 months of radiation therapy
  Patient reported bowel via EPIC-26 (The Expanded Prostate Cancer Index Composite) questionnaire.
To determine whether adaptive SBRT to prostate compared to non adaptive image guided SBRT to prostate results in different rates of patient reported outcomes, acute toxicity. | Within 3 months of radiation therapy
  Patient reported sexual outcomes via EPIC -26 (The Expanded Prostate Cancer Index Composite) questionnaire.
To determine whether adaptive SBRT to prostate compared to non adaptive image guided SBRT to prostate results in different rates of patient reported outcomes, acute toxicity. | Within 3 months of radiation therapy
  Patient reported urinary outcomes via EPIC-26 (The Expanded Prostate Cancer Index Composite) questionnaire.
To determine whether adaptive SBRT to prostate compared to non adaptive image guided SBRT to prostate results in different rates of patient- reported outcomes, acute toxicity. | Within 3 months of radiation therapy
  Patient reported urinary outcomes via I-PSS (International Prostate Symptom Score).
To determine whether adaptive SBRT to prostate compared to non adaptive image guided SBRT to prostate results in different rates of patient- reported outcomes at 2 years, late toxicity. | 2 years following radiation.
  Patient reported bowel, sexual, and urinary outcomes via EPIC-26 (The Expanded Prostate Cancer Index Composite) at 2 years.
To determine whether adaptive SBRT to prostate compared to non adaptive image guided SBRT to prostate results in different rates of patient- reported outcomes at 2 years, late toxicity. | 2 years following radiation
  Patient reported urinary outcomes via I-PSS (International Prostate Symptom Score) questionnaire at 2 years.
To determine whether adaptive SBRT to prostate compared to non adaptive image guided SBRT to prostate results in different cumulative incidence of biochemical failure and distant metastases. | Within 3 months of radiation therapy
  Determine the acute toxicity at 3 months via CTCAE v5.0 (Common Terminology Criteria for Adverse Events).
To determine whether adaptive SBRT to prostate compared to non adaptive image guided SBRT to prostate results in different cumulative incidence of biochemical failure and distant metastases. | 2 years following radiation
  To determine the late toxicity at 2 years via the CTCAE v5.0 (Common Terminology Criteria for Adverse Events).
To determine the economic impact of adaptive SBRT to prostate compared to non adaptive image guided SBRT to prostate. | 2 years following radiation
  The cumulative incidence of biochemical failure and distant metastases, economic impact.

OTHER OUTCOMES:
To determine the impact of magnetic resonance-based adaptive SBRT (e.g., MR-Linac) versus CT-based adapted SBRT (e.g., Ethos) across each of the primary and secondary objectives. | within 2 years following radiation
  MR-based vs CT-based adaptive SBRT across each of the primary and secondary endpoints.
Tertiary endpoints: To determine whether cumulative dosimetric differences between adaptive and non adaptive prostate SBRT correlate with each of the primary and secondary objectives. | within 2 years following radiation
  Adaptive vs non-adaptive target and organ-at-risk dosimetric differences.

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Center, Toronto, Ontario, Canada